CLINICAL TRIAL: NCT07270913
Title: The Effect of a Gender Education Program Based on the Com-B Model Developed for Newlywed Couples and Home Monitoring on Individuals and Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selma Kahraman (Other)
Responsible Party: Sponsor-Investigator, Selma Kahraman, Professor Doctor, Harran University
Organization: Harran University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Date:11.13.2025, No: 2025/354
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Newly Married Couples; Gender Equality; COM_B Model; Home Monitoring Follow-up; Family Dynamics; Education
Keywords: Gender; COM-B Model; Behavior Change; Newly married couples; Family Health; Home monitoring; Family harmony
MeSH Terms: conditions — Coitus | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gender education and home monitoring (Experimental)
  Interventions: Behavioral: information
- 2. Control (No Intervention)

INTERVENTIONS:
Behavioral: information — COM-B Gender İnformation
  Other Names: Home monitoring
  Arms: Gender education and home monitoring

SUMMARY:
Introduction and Aims:

The family, recognized as the smallest and most powerful social unit that forms society, is an arena where gender roles, gender identities, and inequalities are reproduced and developed. The establishment, maintenance, and continuation of a healthy marriage is the source of healthy families and, naturally, healthy individuals. Therefore, research on newly married individuals is valuable as it sheds light on future generations. This research began with the question, "How should effective gender education be designed to minimize gender inequality and the problems arising from it?" This research presents a study protocol to evaluate the effectiveness of a gender education program based on the Capacity, Opportunity, and Motivation to Behave (COM-B) model. Furthermore, this study aims to take solid steps in the first stage of family formation through a one-year follow-up of newly married couples and thus create healthy and strong families.

Method:

This study will be conducted as a two-phase, prospective, single-center, two-group (1:1) parallel design, pre-test-post-test randomized controlled trial. The Capacity, Opportunity, and Motivation Behavior (COM-B) model is a theoretical framework consisting of six components to understand and support behavior change. In the first phase, a gender education program based on the COM-B model (COMBTC) will be developed, and in the second phase, the effectiveness of COMBTC will be evaluated with 100 newly married couples. The sample will consist of 100 couples who have been married for no more than one month and live in central Şanlıurfa, divided into intervention and control groups at a 1:1 ratio. Participants in the intervention group will undergo a 3-week, multi-component education program based on the COM-B model, while participants in the control group will receive routine general advice. Assessments will be conducted at baseline, after the education, and at 6-11 months. Research data will be collected using a personal information form, a healthy family scale, a marital role expectations scale, a marital problem-solving scale, and a family harmony scale. The data will be evaluated using descriptive statistical analyses and relevant tests.

DETAILED DESCRIPTION:
Gender-based issues typically manifest as discrimination and equity problems rooted in the different roles and stereotypes that society imposes on women and men. There is ample evidence that gender inequalities and restrictive norms negatively impact health; however, far fewer studies have focused on testing solutions. Identifying individuals' attitudes toward gender equality and potential sexist attitudes and behaviors is not sufficient on its own. In order for these sexist attitudes and behaviors to transform into more egalitarian attitudes, educational programs on gender equality must be designed, implemented, and their effects determined. This is because education is the best tool for bringing about and sustaining change in relation to gender equality. Education has a significant impact on individuals' awareness of gender inequalities in society, the formation of social consciousness regarding gender equality, and ensuring the continuation of this egalitarian structure in democratic societies. Discussions on gender education are intense but fragmented. Therefore, the aim of this research is to conduct a needs analysis regarding the level and content of gender education and to develop recommendations on the level and content of effective education.

In today's society, where divorces and unhappy marriages are rapidly increasing, healthy marriages are more difficult to achieve than in the past. The main reason for this is that societies undergoing rapid change are under pressure from modernism, weakening traditional structures and preventing new behavioral patterns from taking root. In our time, building strong families through healthy marriages has become much more important. The more solid and healthy the foundations of a family are within a community, the more solid and healthy the society formed by that family will be. Healthy generations are raised in a family environment. For this reason, this project focuses on newly married couples who are just starting to build a family. Gender education for newly married individuals, who are at the forefront of the family where gender roles are first observed and gender identities and inequalities are reproduced and developed, plays an important role in overcoming gender-related problems. This study focus on newly married couples, i.e., young people or young adults, also highlights the global opportunity to address gender-based constraints on health and well-being at an early age to ensure that young people benefit from their effects throughout their lives and offers the opportunity to prevent gender-based health inequalities through early intervention. Interventions targeting gender roles in newly married couples continue, but very few address the underlying causes expected for the intervention to be the underlying behavioral change mechanisms expected for the intervention to be effective. To increase the effectiveness of the intervention, new tools in behavioral science, such as the COM-B model (competence, opportunity, motivation, and behavior), have been used to understand behaviors in intervention development.

The main purpose of the COM-B model is to determine what needs to change to create behavioral change and what needs to be done. Behavioral change requires understanding the factors that drive behavior. To address this, researchers Michie and colleagues developed a model called the COM-B model. According to this model, for behavioral change to occur, the individual must have sufficient ability and opportunity, and their motivation must increase (West and Michie, 2020). In the model, to create behavioral change, individuals' abilities and opportunities are identified, their motivation is increased, and behavioral change is created. In the model, ability includes the physical and psychological capacity that the individual possesses to perform the behavior. Opportunity encompasses the physical and social factors that influence an individual's ability to perform the behavior. Motivation is a process that involves the individual's decision-making and implementation for the behavior to occur (West and Michie, 2020; Ögel and Şimşek, 2023). There are nine intervention initiatives around the center to implement the model: education, persuasion, encouragement, coercion, instruction, restrictions, environmental restructuring, modeling, and activation. Education ensures that the person's level of knowledge is increased. Persuasion is the use of communication to change the person's feelings about the behavior and to bring about behavioral change. Incentives reward the person for behavioral change. Pressure creates the expectation of punishment or penalty. Restrictions involve using rules to create change in the target behavior. Environmental restructuring involves changing the physical and social environment. Instruction involves acquiring and developing skills. Modeling provides a situation for the person to imitate or take as an example. Enabling refers to initiatives that reduce barriers by increasing skills and opportunities. Therefore, the COM-B model can provide a systematic framework for designing and implementing gender education interventions in newly married individuals to increase the effectiveness of intervention programs. This is because there is a lack of evidence on instilling and implementing egalitarian gender roles in newly married individuals, and research is needed to apply the COM-B model to objectively reflect its impact. In this study, numerous strategies and techniques will also be designed and adapted to optimize the gender education program and provide practical evidence, guided by this theoretical model.Improving quality in public health practices is possible by facilitating behavioral change in individuals (Michie et al., 2011). Controlling unhealthy behaviors is considered the ultimate goal of health professionals working in this field. The best way to achieve this goal is to provide services that comprehensively assess the individual's environment and surroundings. One such service is home visits. This is because home visits enable the creation of healthy communities and the provision of comprehensive healthcare in many areas to individuals, families, and community groups. Therefore, home visits are an important initiative in terms of monitoring couples in their environment, addressing all factors, observing mistakes made, and intervening immediately.

ELIGIBILITY:
Inclusion Criteria:

* Married 1 month ago
* The woman and her husband are literate in Turkish
* Being a housewife
* Growing up in Şanlıurfa and residing in the center
* Authorizing participation.

Exclusion Criteria:

* - Married for more than 1 month or single
* Being a working woman
* Not knowing Turkish
* Not living in the center of Şanlıurfa
* Currently participating in any other intervention program

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To ensure the formation of egalitarian role expectations in marriage | First 2 months of preparation and education Through study completion, an average of 10 month
  Change From Baseline in healthy family scale at 10 month. Change From Baseline in marital role expectations scale at 10 month. Change From Baseline in marital problem-solving scale at 10 month Change From Baseline in family harmony at 10 month
Ensuring the formation of egalitarian role expectations in marriage | 10 month
  Research data will be collected using a personal information form, a healthy family scale, a marital role expectations scale, a marital problem-solving scale, and a family harmony scale.

IPD SHARING:
Plan to Share IPD: Undecided